CLINICAL TRIAL: NCT07241026
Title: The Impact of Mental Rotation and 3D Perception Abilities on the Development of Practical Skills in Physiotherapy and Rehabilitation Students
Brief Title: Mental Rotation, 3D Perception, and Practical Skill Development in Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assc. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AIBU-FTR-RK-13
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Educational Problems
Keywords: Mental Rotation; Physiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective parallel group with double-blinded design
Who Masked: Participant, Outcomes Assessor
Masking Description: Control group will receive sham mental rotation and 3D perception exercises fand outcome assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D spatial cognition training and mental rotation (Experimental): Participants will receive a structured mental rotation and 3D spatial cognition training program, consisting of immersive virtual reality (VR) practice, computerized rotation tasks, and hands-on spatial exercises
  Interventions: Other: Spatial-Cognitive & 3D-Perception Training Program
- Sham 3D spatial cognition training and mental rotation (Sham Comparator): Participants will receive a sham mental rotation and 3D spatial cognition program, consisting of non-spatial computerized tasks and general educational activities without targeted spatial training
  Interventions: Other: Sham Spatial-Cognitive & 3D-Perception Training Program

INTERVENTIONS:
Other: Spatial-Cognitive & 3D-Perception Training Program — Participants will undergo a 60-minute training session, consisting of immersive 3D/VR practice, computerized mental rotation tasks, and hands-on spatial exercises. Each session will begin with a 20-minute VR-based activity in which students interact with anatomical models and 3D objects, rotating and orienting them to match different views and cross-sections. This will be followed by a 20-minute computerized module, where participants complete adaptive mental rotation tasks of varying angular disparity, including both object-based and body-posture items. The final 15-20 minutes will include practical spatial exercises, such as assembling 3D anatomical puzzles, reach-and-place tasks, and proprioceptive orientation drills.Training will be delivered 3 days per week for 8 weeks.
  Arms: 3D spatial cognition training and mental rotation
Other: Sham Spatial-Cognitive & 3D-Perception Training Program — Participants will undergo a 60-minute training session, consisting of non-spatial computerized tasks, general cognitive exercises, and low-demand hands-on activities. Each session will begin with a 20-minute computer-based activity presenting neutral content, such as quizzes, word puzzles, or simple problem-solving tasks, without requiring 3D manipulation or mental rotation. This will be followed by a 20-minute module of general cognitive tasks, including memory or attention exercises unrelated to spatial orientation. The final 15-20 minutes will include low-intensity hands-on activities, such as organizing materials or following simple step-by-step instructions, designed to match the duration and engagement of the intervention arm without targeting spatial cognition. Training will be delivered 3 days per week for 8 weeks.
  Arms: Sham 3D spatial cognition training and mental rotation

SUMMARY:
This study investigates the role of mental rotation and 3D perception abilities in shaping the practical skill performance of physiotherapy and rehabilitation students. By exploring the relationship between spatial cognitive abilities and hands-on competencies, the research aims to provide insights that may improve educational strategies and clinical training outcomes.

DETAILED DESCRIPTION:
Practical skills are fundamental to physiotherapy and rehabilitation education, requiring students to accurately interpret anatomical structures, movement patterns, and therapeutic techniques in three-dimensional space. Cognitive abilities such as mental rotation and 3D perception are considered essential in processing spatial information and transferring theoretical knowledge into clinical practice. However, limited research has explored how these spatial abilities influence the acquisition and execution of practical competencies in physiotherapy training.

This study aims to assess the relationship between mental rotation ability, 3D spatial perception, and the practical performance of physiotherapy and rehabilitation students. Standardized spatial ability tests will be used alongside practical skill assessments to identify correlations between cognitive factors and clinical task execution. The findings are expected to contribute to curriculum design by highlighting the importance of integrating spatial training modules and potentially guiding student selection or tailored support strategies.

The aim of this study is to examine the impact of mental rotation and 3D perception abilities on the development and performance of practical skills in physiotherapy and rehabilitation students, with the goal of enhancing educational methods and optimizing clinical training outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and provide written informed consent
* Normal or corrected-to-normal vision

Exclusion Criteria:

* History of neurological or musculoskeletal disorders affecting upper-limb function or spatial cognition
* Severe visual impairments that cannot be corrected
* History of epilepsy, severe motion sickness, or vestibular disorders
* Participation in other spatial-cognition or VR-based training programs within the last 6 months
* Use of medications affecting cognitive function or balance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Grade Point Average (GPA) | Baseline, eight weeks and 48 months
  To evaluate the overall academic performance of participants, Grade Point Average (GPA) will be collected from university records. GPA is calculated on a 4.0 scale, with 0.0 representing failing performance and 4.0 representing excellent academic achievement. Higher scores indicate better academic performance.
Purdue Spatial Visualization Test: Rotations (PSVT-R) | Baseline, eight weeks and 48 months
  To assess participants' spatial visualization and mental rotation abilities, the PSVT-R will be administered. The test comprises 30 multiple-choice items, each with a single correct answer, scored 1 for correct and 0 for incorrect responses. Total scores range from 0 to 30, with higher scores reflecting stronger spatial visualization skills.

SECONDARY OUTCOMES:
Corsi Block-Tapping Test | Baseline and eight weeks
  Involves mimicking a sequence of up to nine spatially separated blocks tapped by the examiner. The length of the longest sequence correctly recalled is the score. Higher scores indicates better spatial abilities
Test Anxiety Inventory | Baseline and eight weeks
  To examine whether there is a change in the level of anxiety experienced by students during the exam, a 5-question short version of Test Anxiety Inventory will be used. The test includes sections related to ease, comfort associated with learning, and alignment of exam questions with the course.
Enjoyment and Recommendation | Baseline and eight weeks
  Participants will fill out a feedback questionnaire regarding the learning instruments using visual analogue scale (0-100mm).
Test Taking Motivation Questionnaire | Baseline and eight weeks
  To assess the level of motivation students exhibit during examinations, the Test Taking Motivation Questionnaire (TTMQ) will be administered. The questionnaire includes items evaluating students' effort, engagement, persistence, and goal orientation during test situations. Each item is rated on a Likert scale, and total scores generally range from 0 to 100, with higher scores indicating greater motivation and engagement in test-taking activities.
Mental Rotation Test | Baseline and eight weeks
  To evaluate the ability to mentally rotate three-dimensional objects, the Mental Rotation Test will be used. The test includes 24 items, each with two correct answers. Each correct response is awarded 1 point, resulting in a total score ranging from 0 to 24. Higher scores indicate greater proficiency in mental rotation tasks.
Puzzle Assembly | Baseline and eight weeks
  Participants were asked to complete 3d printed puzzle of bone fractures and completion time was tracked.
CarMen-Q | Baseline and eight weeks
  Participants were asked to complete the CARMEN-Q (Cognitive Load, Motivation, and Emotion Questionnaire) to evaluate their perceived cognitive load and related psychological responses. The scale includes four subscales: Intrinsic Load, Extraneous Load, Germane Load, and Affective-Motivational Factors (Motivation, Emotion, and Self-Efficacy). Each item is rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores on the cognitive load subscales reflect greater perceived mental effort, while higher scores on motivation, emotion, and self-efficacy indicate more positive learner engagement and affective response.

CONTACTS AND LOCATIONS:
Overall Officials: ramazan kurul, phd, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The dataset can be obtained from the principal investigator upon any reasonable request.
Supporting Information: Study Protocol
Time Frame: After publication of the research.
Access Criteria: ramazankurul@ibu.edu.tr